CLINICAL TRIAL: NCT02450825
Title: Comparison of Three Scores for Ultrasound Assessment and Monitoring of Pulmonary Aeration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15.012
Record Dates: First submitted 2015-05-12; First posted 2015-05-21 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Atelectasis; Pneumonia; Acute Respiratory Distress Syndrome; Pulmonary Embolism; Hypoxemia; Dyspnea
MeSH Terms: conditions — Pulmonary Atelectasis; Pneumonia; Respiratory Distress Syndrome; Pulmonary Embolism; Hypoxia; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mechanically ventilated patients (Other): Mechanically ventilated patients who underwent a computed tomographic scan for dyspnea or hypoxemia will undergo a standardized lung ultrasound examination on Day 1 and Day 2 to 4. The GE Vivid ultrasound system will be used to perform the lung ultrasound examination.
  Interventions: Procedure: Lung ultrasound examination on Day 1 and Day 2 to 4; Device: GE Vivid Ultrasound system
- Spontaneously breathing patients (Other): Spontaneously breathing patients who underwent a computed tomographic scan for dyspnea or hypoxemia will undergo a standardized lung ultrasound examination on Day 1 only. The GE Vivid ultrasound system will be used to perform the lung ultrasound examination.
  Interventions: Procedure: Lung ultrasound examination on Day 1; Device: GE Vivid Ultrasound system

INTERVENTIONS:
Procedure: Lung ultrasound examination on Day 1 and Day 2 to 4 — A standardized lung ultrasound examination using the GE Vivid ultrasound system will be performed following the tomographic scan on Day 1 and repeated on Day 2 to 4. Correlation of ultrasound-based aeration scores will be done with lung aeration measured by computed tomographic images.
  Arms: Mechanically ventilated patients
Procedure: Lung ultrasound examination on Day 1 — A standardized lung ultrasound examination using the GE Vivid ultrasound system will be performed following the tomographic scan on Day 1 only. Correlation of ultrasound-based aeration scores will be done with lung aeration measured by computed tomographic images.
  Arms: Spontaneously breathing patients
Device: GE Vivid Ultrasound system — The GE Vivid ultrasound system will be used for all lung ultrasound examinations performed in this study.

SUMMARY:
This study is designed to compare three ultrasound-based aeration scores that were previously validated in specific populations, and to assess their correlation with computed tomographic measurement of pulmonary aeration in a population with different pathologies.

Hypothesis: The "Loss of Aeration Score" will be more accurate than a simplified version and another widely used score, the "Lung Ultrasound Score".

DETAILED DESCRIPTION:
Assessment of lung aeration may have a great impact in the management of mechanical ventilation and follow-up of diverse lung pathologies. Computed tomographic scan is the gold standard method of lung aeration measurement but is rarely used because it requires transport of critically ill patients end exposes them to radiations. For these reasons, lung ultrasound would be an attractive alternative. Variants of different ultrasound-based aeration scores have been validated in different specific populations, but there is no comparison study that defines the more accurate score that should be used in a population with different pathologies.

Methods: Patients undergoing a computed tomographic scan for dyspnea or hypoxemia will have a standardized lung ultrasound examination on Day 1. For mechanically ventilated patients only, a lung ultrasound examination will be repeated on Day 2 to 4. End expiratory lung volume will also be measured in mechanically ventilated patients on Day 1 and Day 2 to 4. Lung ultrasound images will be interpreted blindly. Correlation of ultrasound-based aeration scores will be done with lung aeration measured by computed tomographic images.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized or visiting the emergency room
* Will undergo a computed tomographic scan for dyspnea or hypoxemia

Exclusion Criteria:

* Poor echogenicity (morbid obesity, multiple thoracic dressings)
* Contraindications to superior limbs or torso mobilization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Correlation of ultrasound-based aeration scores with computed tomographic measurement of pulmonary aeration. | Day 1

SECONDARY OUTCOMES:
Correlation of ultrasound-based aeration scores and expiratory lung volume variation. | Day 2 to Day 4
  In mechanically ventilated patients, correlation of ultrasound-based aeration scores and expiratory lung volume variation between Day 1 and Day 2 to 4 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No